CLINICAL TRIAL: NCT06957509
Title: Salivary Metaproteome as a Prediction Tool in Early Childhood Caries
Brief Title: Analysis of Salivary Proteins in Young Children as an Device to Improve Caries Risk Assessment
Acronym: DecodECC
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Folktandvården Stockholms län AB (Other Government)
Responsible Party: Principal Investigator, Franziska Hetrodt, Lecturer, Karolinska Institutet
Other Study IDs: 2024-07097-01
Record Dates: First submitted 2025-04-02; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Early Childhood Caries (ECC)
Keywords: early childhood caries; saliva; metaproteins; caries risk assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- NC: caries-free children
- C: children with clinically detectable caries (initial or manifest)
- proteom Järva: proteome of 3-year-old children examined in Folktandvården Järva
- proteom Danderyd: proteome of 3-year-old children examined in Folktandvården Danderyd

SUMMARY:
The goal of this observational study is to learn if the composition of salivary proteins in 3-year-old children, from communities with documented varying caries risks, can be used to identify future diagnostic predictors for caries risk.

The main question to answer is:

• Can the host´s salivary protein profile (expression and abundance) show a correlation with the caries prevalence between the individuals in the different study cohorts?

Two cohorts of children with different documented demographic characteristics in the region of Stockholm (Sweden) will be examined.

Participants will be asked to provide saliva samples and undergo clinical oral examinations conducted by trained dental practitioners.

DETAILED DESCRIPTION:
Project summary

The term early childhood caries (ECC) describes the presence of one or more decayed, missing (due to caries) or filled primary teeth in children aged six years or younger. It has been shown that risk factors for ECC are frequent sugar consumption, inadequate oral hygiene as well as the colonization with cariogenic bacteria, such as the group of mutans streptococci, which are considered to be the main etiological agents of tooth decay in children. Other bacteria, such as Prevotella spp. and Lactobacillus spp., as well as fungus Candida albicans, were shown to be associated to the development and progression of ECC. Proteins in human saliva can influence the viability of oral microorganisms by various innate defense mechanisms, thus affect the composition of the oral microflora. Simultaneously bacteria are producing proteins to enhance various processes, e.g., the production of polysaccharides. While the word proteomics covers the exploration of all proteins from one species, metaproteomics relates to the investigation of proteins from microbial communities in interaction with the host, e.g. the host-microbiota crosstalk. Overall, the protein composition in young children's saliva, be it of microbial or human origin, could assist in biomarker implementation for early diagnosis as well as risk assessment of ECC.

This study aims to explore the overall salivary protein composition in cohorts of 3-year-old children from Swedish communities of varying risk for ECC, using high-throughput proteomics.

In brief, 50 3-year-old children will be recruited at two Public Dental Healthcare Centers, Folktandvården Danderyd and Folktandvården Järva, respectively. The project is structured in a clinical part (stage 1) and an analytical laboratory part (stage 2). Stage 1 will entail the recruitment of patients, the collection of saliva swab samples as well as the clinical examination, with particular emphasis on the presence of ECC. Stage 2 comprises the molecular analytical part during which the proteomic characterization of the saliva will take place. This molecular analytical part will be performed at the Department of Dental Medicine at Karolinska Institutet, with the support of the respective core facilities (Scaleless).

The investigators hypothesize that there are differential host proteomic and metaproteomic salivary profiles in ECC-affected children compared to caries-free children, and that these are associated with already identified risks for ECC posed between the two community-distinct cohorts.

Purpose and aim

This project aims to utilize proteomic technologies for analyzing the composition of the saliva in two 3-year-old children cohorts from communities with documented varying caries risks, with the purpose of identifying future molecular diagnostic risk- and health-promoting factors for ECC.

Primary Research Questions

• Can the host's proteome and metaproteome profile (protein expression and abundance) show a correlation with caries prevalence among individuals in the different cohorts in the study?

Secondary Research Questions

1. How does the caries profile differ between the recruited child cohorts from different socioeconomically characterized communities in Stockholm?
2. How does the host's proteome and metaproteome profile differ between caries-affected and caries-free children?
3. How does the host's proteome and metaproteome profile correlate with:

   * a) Risk factors addressed in interview questionnaires?
   * b) The clinical status and severity of caries prevalence?

The investigators hypothesize that a higher prevalence of ECC will be registered at the Folktandvården Järva, compared to Folktandvården Danderyd and that there will be proteome (host and microbial) variations in the salivary composition according to clinical and socioeconomic risk statuses.

Background

Early childhood caries (ECC) is defined as caries found in the primary dentition of preschool-aged children, i.e. children younger than 6 years of age. Even though significant advancements were shown in preventive dentistry, ECC remains a major health issue for many children worldwide. Despite limited representative data, reports from various countries show that the prevalence of ECC in children aged 2-3 years generally ranges from 12% - 27% . It has been shown that ECC is likely to be found more prevalent in socially disadvantaged minority groups with lower income. Previous studies performed in areas with high risk for dental caries in Stockholm indicate that an immigrant background, considering factors like culture, ethnicity, lifestyle, dietary pattern, and oral hygiene practices, is a strong predictor for the development of ECC. This leads to the hypothesis that differences in the cariological status may be found in socioeconomically different communities of the County of Stockholm, such as the Danderyd and Järva communities.

Furthermore, saliva has been discussed as a crucial biological modulator, involved in the maintenance of oral health. Based on the simplicity and noninvasiveness of saliva sample collection, there has been recently an increasing interest in the usage of this complex body fluid as a diagnostic tool.

Several studies have explored the potential use of salivary proteins as biomarkers for caries frequency and suggested correlations between both the total concentration as well as the nature of salivary proteins and the occurrence of dental caries.

Additionally, a strong correlation has been found between higher levels of microbials, such as mutans streptococci, Prevotella spp., and C. albicans, and increased caries prevalence in preschool children. While the term proteomics involves the study of all proteins from a single species, mass spectrometry-based metaproteomics focuses on characterizing proteins of bacterial communities in interaction with the host. In the literature, only a limited number of studies have addressed the metaproteome of dental caries in biofilms.

However, these findings have typically been observed in adolescents or adults, and investigations of the interactions between the oral microbiome and the host immune system in young children are lacking.

Thus, this study aims to expand the knowledge of human and bacterial metaproteomic characteristics to implement potential biomarkers for ECC, aiding in prevention, risk assessment, and therapy for ECC.

Project description

This cross-disciplinary project will be accomplished through the collaboration between Folktandvården at Stockholm's läns landstinget (SLL) (Dr. Maria Anderson) and the Department of Dental Medicine (KI) (Dr. Franziska Hetrodt and Prof. Georgios Belibasakis). Furthermore, the analytical part of the project will be supported by the Proteomics Biomedicum facility at KI Campus Solna. This project will be performed within a clinical (stage 1) and a laboratory part (stage 2). The proteomics workflow will be performed according to established protocols.

Stage 1. Recruitment, clinical examination, and saliva sample collection A power analysis, based on a two-tailed F test of variance for two-group comparison (proteome 3-year-old children examined in Folktandvården Danderyd vs 3-year-old children examined in Folktandvården Järva), with a minimum effect size of 2 (log2-fold changes), a minimum power of 80%, a significance level of 5%, and a 10% excess to account for potential dropouts or incomplete data, revealed a minimum sample size of 50 participants being required in both study groups.

Children with or without ECC will be recruited from the Folktandvården clinic in Järva and Danderyd. In Sweden dental healthcare is free of charge for children, and the first dental examination of the oral health status is routinely performed at the age of three years. For this reason, the Folktandvården clinics in Stockholm arrange events evaluating the oral health status of 3-year-old infants. This is a unique opportunity to gather and examine on one occasion large community groups of children with the same age, as well as comparable environmental and socio-economic factors.

The investigators are therefore aiming for two study cohorts consisting of self-defined populations with calibrated date and time. The recruitment of the two study cohorts will be monitored by Dr. Maria Anderson and Dr. Franziska Hetrodt. Written informed consent will be obtained as prerequisite for study participation. Medical history will be taken and children with caries-affected diseases, e.g. asthma, will be registered. Demographic information such as sex will be recorded for each study participant. Information about general diseases, eating and tooth brushing habits as well as socio-cultural factors, such as language, ethical background, education level of parents etc. will be recorded by means of a questionnaire.

All patients (n=100) will be requested to abstain from eating, drinking and all oral hygiene procedures for 2 h prior to sampling. Patients will be asked to rinse their mouth with tap water and wait for 5 min to avoid sample dilution. Saliva collection will be performed by the swab-based saliva collection method [SalivaBio Children's Swab (Item No. 5001.06)]. For this, cotton swaps will be gently moved under the tongue, then placed into 15mL sterile sample tubes and immediately refrigerated until transferred to the -80°C freezer for snap-freezing. The time between sample acquisition and freezing should not exceed 30 min to avoid sample damage. A unique ID code will be given to each sample that is linked to the patients' record. Before the analysis, saliva samples were thawed on ice, centrifuged (4000 rpm, 20 min, 4 °C) to obtain saliva supernatants, and frozen at -80 °C again until further use. Clinical standard examination of each individual child will be conducted after acquisition of saliva samples by calibrated examiners (dentists or dental oral hygienists). Calibration will be performed with clinical videos and instructions prior to study member recruitment. Caries frequency will be registered by the decayed missed filled teeth (dmft) index and ICDAS merged. Dental treatment will be performed as indicated. The saliva collection as well as dental evaluation and risk classification in the patient journal T4 (Carestream Dental) is performed by employees of Folktandvården in Stockholm.

Stage 2. Proteome profiling of the collected saliva samples The high throughput proteomics analyses performed in this project includes both host proteomics (human proteins) and metaproteomics (polymicrobial community proteins). These analyses need the combination of the expertise and facilities provided at the ANA Futura laboratories at Campus Flemingsberg and the Proteomics Biomedicum facility at Campus Solna. Saliva samples will be pre-handled and then processed through a label-free quantitative proteomic analysis. The protein concentration of the samples will be measured and then diluted to the same amount (typically 20 µg/reaction). For mass spectrometric single-cell proteomics analysis, single cells in 96-well plates will be send to the Proteomics Biomedicum facility at Campus Solna and analyzed in service mode according to established routines. In brief, the samples will first undergo protein extraction and trypsin-digest. Thereafter, peptide samples will be labelled using tandem mass tag (TMT) reagents, dried and then subjected to liquid chromatography with tandem mass spectrometry (LC-MS/MS) analysis. The acquired proteome data will then be annotated against known protein databases, and the protein regulation patterns and pathway enrichments between the different study groups will be assessed.

General timeline

This is a 3 year-project according to the following steps. The ethical application was approved during fall 2024 and the clinical part (stage 1) entailing the participant recruitment and sample collection is planned for spring 2025. The laboratory part (stage 2) including salivary analysis will be initiated after the completion of stage 1 (fall 2025 - fall 2026) to ensure equal processing of all samples. Data analysis will be conducted, and findings will be published in fall 2027.

Significance

Early childhood caries is a major oral health problem, affecting infants and preschool children worldwide. The main risk factors in the formation of ECC can be categorized as microbiological, dietary, and environmental risk factors, as it was previously shown that ECC occurs mainly in socially disadvantaged populations. When diagnosed with ECC, children will likely exhibit a more advanced clinical picture of the disease in the future. So far, the role of molecular mechanisms and the host-microbiota crosstalk in caries-active vs. caries-free children, are not fully understood. The findings of this project will contribute to a better understanding of the appearance of molecular ways and help eventually to identify potential therapeutic targets and biomarkers for diagnosis and prevention before the clinical manifestation of the disease occurs. In addition, potential salutogenic biomarkers could be found for children exposed to a vulnerable environment, but surviving caries-free.

ELIGIBILITY:
Inclusion Criteria:

* 3-year-old children residing in the areas served by Folktandvården Danderyd and Järva, respectively
* Written consent, signed by both parents (guardians)

Exclusion Criteria:

* children older than three years
* medication intake, and antibiotic use at the time of examination
* children who have consumed food, drink, or used oral hygiene products within 2 hours before the dental visit
* children who appear uncooperative during saliva sampling

Ages: 3 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children will be recruited in conjunction with their mandatory three-year examination at two of Folktandvården's clinics: Järva (care need area 3-4) and Danderyd (care need area 1-2). Dental care is free for children, and the first oral health status examination by a dentist is routinely performed when the child turns three years old. Therefore, Folktandvården's clinics in Stockholm organize events (3-year-old parties) where the first examination of 3-year-old children is conducted. This is a unique opportunity to simultaneously call in and examine community groups of children of the same age, with comparable environmental and socioeconomic factors. We are therefore aiming for two study cohorts consisting of self-defined populations with calibrated age.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Differential protein expression across caries severity levels | up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Folktandvården Stockholms län AB, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruan W, Sun C, Gao Q, Shrivastava N. Metaproteomics associated with severe early childhood caries highlights the differences in salivary proteins. Arch Oral Biol. 2021 Nov;131:105220. doi: 10.1016/j.archoralbio.2021.105220. Epub 2021 Jul 29. PMID 34461447
- [Background] Belda-Ferre P, Williamson J, Simon-Soro A, Artacho A, Jensen ON, Mira A. The human oral metaproteome reveals potential biomarkers for caries disease. Proteomics. 2015 Oct;15(20):3497-507. doi: 10.1002/pmic.201400600. Epub 2015 Sep 22. PMID 26272225
- [Background] Paes Leme AF, Bellato CM, Bedi G, Cury AA, Koo H, Cury JA. Effects of sucrose on the extracellular matrix of plaque-like biofilm formed in vivo, studied by proteomic analysis. Caries Res. 2008;42(6):435-43. doi: 10.1159/000159607. Epub 2008 Oct 3. PMID 18832830
- [Background] Ahmad P, Hussain A, Carrasco-Labra A, Siqueira WL. Salivary Proteins as Dental Caries Biomarkers: A Systematic Review. Caries Res. 2022;56(4):385-398. doi: 10.1159/000526942. Epub 2022 Sep 20. PMID 36116431
- [Background] Anderson M, Dahllof G, Warnqvist A, Grindefjord M. Development of dental caries and risk factors between 1 and 7 years of age in areas of high risk for dental caries in Stockholm, Sweden. Eur Arch Paediatr Dent. 2021 Oct;22(5):947-957. doi: 10.1007/s40368-021-00642-1. Epub 2021 Jun 9. PMID 34106458
- [Background] Hemadi AS, Huang R, Zhou Y, Zou J. Salivary proteins and microbiota as biomarkers for early childhood caries risk assessment. Int J Oral Sci. 2017 Nov 10;9(11):e1. doi: 10.1038/ijos.2017.35. PMID 29125139
- [Background] Bostanci N, Selevsek N, Wolski W, Grossmann J, Bao K, Wahlander A, Trachsel C, Schlapbach R, Ozturk VO, Afacan B, Emingil G, Belibasakis GN. Targeted Proteomics Guided by Label-free Quantitative Proteome Analysis in Saliva Reveal Transition Signatures from Health to Periodontal Disease. Mol Cell Proteomics. 2018 Jul;17(7):1392-1409. doi: 10.1074/mcp.RA118.000718. Epub 2018 Apr 2. PMID 29610270
- [Background] Vegvari A. Mass Spectrometry-Based Analytical Strategy for Single-Cell Proteomics. Methods Mol Biol. 2022;2420:63-72. doi: 10.1007/978-1-0716-1936-0_6. PMID 34905166